CLINICAL TRIAL: NCT02643355
Title: Utility of Olanzapine in the Treatment of Opioid Withdrawal in the Emergency Department
Brief Title: Utility of Olanzapine in the Treatment of Opioid Withdrawal in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR# 15-4004
Record Dates: First submitted 2015-12-17; First posted 2015-12-31 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Narcotic Withdrawal; Opiate Withdrawal; Emergency Department
MeSH Terms: conditions — Substance Withdrawal Syndrome; Emergencies | interventions — Olanzapine; Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care - Olanzapine (Experimental): Drug of interest in the study - Olanzapine
  Interventions: Drug: Olanzapine
- Standard of Care - Clonidine (Active Comparator): Standard of care - clonidine
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Olanzapine
  Arms: Standard of Care - Olanzapine
Drug: Clonidine
  Arms: Standard of Care - Clonidine

SUMMARY:
Withdrawal from opioids is a clinical scenario that emergency department physicians encounter frequently. Patients who present with opioid withdrawal display symptoms such as agitation, anxiety, myalgias, abdominal pain, diarrhea, nausea, and vomiting. Currently, the standard treatment for opioid withdrawal is clonidine (an alpha-2 adrenergic agonist), as well as supportive cares (anti-emetics, intravenous fluids). Olanzapine is an atypical antipsychotic that is given frequently in the ED for many of the same symptoms that are seen in patients who are experiencing opioid withdrawal, however its use in this toxidrome has never been studied. The hypothesis of this study is that olanzapine is a safe and efficacious option when compared to clonidine for the treatment of opioid withdrawal in the emergency department.

DETAILED DESCRIPTION:
This study will be a randomized control trial where patients will be randomized to receive intramuscular olanzapine or oral clonidine as the first intervention given for treatment of opiate withdrawal. This study will not be blinded.

Screening and enrollment: Research Associates will screen patients by review of the electronic medical record. When these patients are identified, the RA will approach the CITI trained ED provider who will obtain written informed consent. Allergies to either medication will be screened for in Epic by the research associates. Allergies will also be verified by the provider who is completing the consent.

Study protocol: If the patient consents to enroll in the study, the research associate will randomize the patient to receive olanzapine or clonidine as the first treatment intervention. The ED provider will then order that medication for the patient and will it be administered by nursing staff. At this time the provider may order the patient to have a peripheral IV placed and IV fluids administered at their discretion. No other supportive measures (anti-emetics, non-narcotic pain medications) may be given at this time.

Prior to medication administration, the research associate will assess the patient's withdrawal symptoms using the Clinical Opiate Withdrawal Scale for withdrawal symptoms. This is a validated tool used to assess degree of withdrawal symptoms by evaluating physiologic and symptomatic parameters. The medical provider will also obtain information regarding the patients opioid use history (what type of opioid used, chronicity of use, date and time of last use). After the study medication administration, patients will be observed for clinical improvement. At 30 minutes, additional medications or interventions may be prescribed at the discretion of the ED provider for symptom control, including crossover of the study medications. The research associate will record which other medications/interventions were ordered, the indication for these interventions, and times administered.

Symptoms will be re-assessed by the research associate using the COWS at 60 minutes, 120 minutes post administration of the initial treatment intervention, as well as at 4 hours post administration (approximately time of discharge from the emergency depatment). At these same time marks, sedation of the patient will be assessed using the overt agitation severity scale (OASS). Throughout the patient's ED stay, the research associate will be monitoring for adverse complications such as allergic reaction, dystonia, akathisia, respiratory complications, or hypotension.

The investigators will conduct preliminary data analysis after the first 25 and 50 patients are enrolled, respectively. Initial power analysis and sample size calculations delineated that the investigators would need 35 patients per arm to detect a 50% difference in the need for rescue medication at 1 hour between the two study medications.

ELIGIBILITY:
Inclusion Criteria:

* Any patients who present to the emergency department where the providers are concerned for opioid withdrawal contributing to their symptoms on presentation is eligible for inclusion.

Exclusion Criteria:

* Age less than 18
* Allergy to either medication (olanzapine, clonidine)
* Inability to give informed consent
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Martel, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the ED only, by ED physicians
Pre-assignment Details: One patient signed consent but withdrew before randomization to drug (Explaining N=70 total)
Groups:
- Olanzapine: Standard of Care Option 1 - Olanzapine
- Clonidine: Standard of Care Option 2 - Clonidine
Period: Overall Study
Arm/Group | Olanzapine | Clonidine
Started | 34 | 35
Completed | 33 | 30
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care - Clonidine: Standard of Care Option 2 - Clonidine
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Standard of Care - Clonidine | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Continuous [Median (Full Range); unit: years] | 35 [22 to 60] | 34 [21 to 67] | 35 [21 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 21 | 15 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 13 | 26
  African-American | 13 | 7 | 20
  Native American | 4 | 5 | 9
  Other | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Received Rescue Medication for Withdrawal Symptoms Within 1 Hour
Description: Rescue Medication (additional medications given for symptoms) within 1 hour of medication administration
Time Frame: 1 Hour
Population: Patients who received medication within 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Clonidine
Number analyzed (Participants) | 33 | 30
Participants | 9 | 19

2. Secondary Outcome: Clinical Opiate Withdrawal Scale Score at 1 Hour Post Medication
Description: Opiate withdrawal scale score for all patients who received medication by one hour
  The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale, ranging from 0 to 48 (5- 12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal).
  This tool can be used to reproducibly rate common signs and symptoms of opiate withdrawal and monitor these symptoms over time. The summed score for the complete scale can be used to help clinicians determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. The 11 items on the scale include scores rate the following symptoms: pulse rate, GI upset, sweating, tremor, restlessness, yawning, pupil size, anxiety, bone or joint aches, gooseflesh skin, runny nose.
Time Frame: At 1 hour
Population: Patients who had COWs score calculated at 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Clonidine
Number analyzed (Participants) | 31 | 27
units on a scale | 5.3 (4.4) | 6.7 (5.0)

3. Secondary Outcome: Clinical Opiate Withdrawal Scale Score at 2 Hours Post Medication
Description: as for outcome 2
Time Frame: 2 hours
Population: Patients who had data available at 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Clonidine
Number analyzed (Participants) | 25 | 22
units on a scale | 4.8 (4.9) | 3.7 (3.5)

4. Secondary Outcome: Clinical Opiate Withdrawal Scale Score at the Time of Disposition
Description: as for outcome 2
Time Frame: Time of Disposition (on average within 6 hours)
Population: Patients who had data available at the time of disposition
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Clonidine
Number analyzed (Participants) | 14 | 13
units on a scale | 4.3 (3.3) | 3.6 (2.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the ED encounter, on average within 6 hours
Description: AEs including hypotension (that resolved without treatment other than fluids), and extrapyramidal side effects are NOT CONSIDERED serious adverse events
Arm/Group | Olanzapine | Clonidine
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 2/33 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=33) | Clonidine (N=30)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0) — dystonic reaction to medication given
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) — akathisia in patient receiving drug
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — blood pressure (systolic) < 90 that resolved without significant treatment (other than IV fluids)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT02643355/Prot_SAP_000.pdf